CLINICAL TRIAL: NCT06197516
Title: Comparison Of Integrated Neuromuscular Inhibition Technique Versus Neuromuscular Reeducation in Patients With Deep Gluteal Syndrome
Brief Title: Comparison Of INIT Versus NMR in Patients With Deep Gluteal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Deep Gluteal Syndrome
Keywords: Trigger point; NMR; INIT; Deep Gluteal Syndrome
MeSH Terms: conditions — Hip socket neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Neuromuscular Inhibition Technique (Experimental): Individuals in Group A, After palpating the trigger point ischemic compression were applied for 20-60 sec while strain counterstain for 60-90 sec and MET is for 7-10 sec. This technique was repeat 3-4 time per session Conventional treatment include Hot Pack for 5mins, AROM exercises ,Home plans include stretching exercise of glutes,hamstring and calf (5-7 reps x 10 sec hold, each).
  Interventions: Other: Integrated Neuromuscular Inhibition Technique
- Neuromuscular Reeducation Technique (Active Comparator): Deep pressure were applied along origin and insertion of Piriformis and hamstring muscle combined with active movement of patient for 5 -15 time as per required (depend upon thickness of scar) per session, 10 sec rest b/w pressure. This technique given 5 time per session. Conventional treatment include Hot Pack for 5mins, AROM exercises ,Home plans include stretching exercise of glutes,hamstring and calf (5-7 reps x 10 sec hold, each).
  Interventions: Other: Neuromuscular Reeducation Technique

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition Technique — After palpating the trigger point ischemic compression were applied for 20-60 sec while strain Counterstain for 60-90 sec and MET is for 7-10 sec.
  Arms: Integrated Neuromuscular Inhibition Technique
Other: Neuromuscular Reeducation Technique — Deep pressure were applied along origin and insertion of Piriformis and hamstring muscle combined with active movement of patient for 5 -15 time as per required
  Arms: Neuromuscular Reeducation Technique

SUMMARY:
Rationale of this research is to evaluate the outcome of Comparison of Integrated Neuromuscular Inhibition technique versus Neuromuscular reeducation on pain in patients with Deep Gluteal Syndrome. The significance of this study is to identify which technique is superior in alleviating the symptoms of deep gluteal syndrome. This study will help gather evidence on the practice of incorporating trigger point therapy in the treatment of deep gluteal syndrome.

DETAILED DESCRIPTION:
Deep gluteal syndrome is a common buttock and posterior hip pain caused by entrapment of the sciatic nerve in the posterior hip region. Nonoperative therapy involves treating the entrapment location, using rest, anti-inflammatories, musclerelaxants, and physical therapy to relieve compression. The purpose of the study was to evaluate the effects of Integrated Neuromuscular Inhibition Technique versus Neuromuscular Reeducation Technique on pain in subject with deep gluteal syndrome. It was a randomized, controlled trial, conducted among deep gluteal syndrome patients. Sample size was 54 by using G Power Tool software. Participantswere randomly assigned to the intervention or control group after a baseline assessment with a lottery ticket and an opaque envelope. All participants in both groups were evaluated on baseline and 12 th Session.

ELIGIBILITY:
Inclusion Criteria:

Both genders Age: 30-50 years Pain due to a non-discogenic sciatic nerve entrapment in the sub gluteal space Pain, tightness and dysesthesias in the buttock area, posterior thigh Buttock pain aggravated with prolong sitting (>20-30 min) Buttock pain aggravated when sitting with limited straight leg raising ability (seated piriformis test) Pain with the passive internal rotation of hip (Freiberg sign) Pain increase in Flexion, Adduction and internal rotation (Positive FAIR test)

Exclusion Criteria:

* Patient with any Intrinsic Etiology such as hemarthrosis, rheumatoid arthritis, infection or gout Patient with any severe trauma, fractures dislocation, subluxation or ligament injury Any pathology or recent injury around the hip, sacroiliac joint, or lumbar spine Limb length discrepancy Recent buttock trauma and bladder/bowel dysfunction

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th week
  Numeric Pain Rate Scale used to assess pain intensity
Goniometer | 4th week
  used to assess lower limb ranges
Lower Extremity Functional scale | 4th week
  LEFS questionnaire have 20 questions will assess the impairment of a patient with lower extremity musculoskeletal condition or disorders
Sciatica Bothersomeness Index | 4th week
  used to measure the participants' level of sciatica. The scale's ratings range from 0 to 24, with higher levels indicating severe sciatica discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Gulberg green campus of Riphah International University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilera-Bohorquez B, Cardozo O, Brugiatti M, Cantor E, Valdivia N. Endoscopic treatment of sciatic nerve entrapment in deep gluteal syndrome: Clinical results. Rev Esp Cir Ortop Traumatol (Engl Ed). 2018 Sep-Oct;62(5):322-327. doi: 10.1016/j.recot.2018.03.004. Epub 2018 May 26. English, Spanish. PMID 29807785
- [Background] Frank RM, Slabaugh MA, Grumet RC, Virkus WW, Bush-Joseph CA, Nho SJ. Posterior hip pain in an athletic population: differential diagnosis and treatment options. Sports Health. 2010 May;2(3):237-46. doi: 10.1177/1941738110366000. PMID 23015944
- [Background] Boyajian-O'Neill LA, McClain RL, Coleman MK, Thomas PP. Diagnosis and management of piriformis syndrome: an osteopathic approach. J Am Osteopath Assoc. 2008 Nov;108(11):657-64. doi: 10.7556/jaoa.2008.108.11.657. PMID 19011229